CLINICAL TRIAL: NCT02061384
Title: A Pilot Trial of 13-cis Retinoic Acid (Isotretinoin) for the Treatment of Men With Oligoasthenoteratozoospermia
Brief Title: RA-2 13-cis Retinoic Acid (Isotretinoin)
Acronym: RA-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, John Amory, Professor, General Internal Medicine, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000564
Record Dates: First submitted 2014-02-10; First posted 2014-02-12 (Estimated); Results first posted 2021-07-30 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-06

CONDITIONS: Male Infertility; Klinefelter's Syndrome; Y-chromosome Microdeletions
Keywords: Infertility
MeSH Terms: conditions — Infertility, Male; Klinefelter Syndrome; Male sterility due to Y-chromosome deletions; Infertility | interventions — Isotretinoin; Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 13-cis retinoic acid (Experimental): 20mg 13-cis retinoic acid twice daily (BID) with meals for 20 weeks
  Interventions: Drug: 13-cis retinoic acid
- Calcitriol 0.25 mcg (Experimental): oral calcitriol 025 mcg BID subjects 11-20 for 20 weeks
  Interventions: Drug: 13-cis retinoic acid; Drug: Calcitriol

INTERVENTIONS:
Drug: 13-cis retinoic acid — Accutane is used for the treatment of severe acne
  Other Names: Accutane; Isotretinoin
Drug: Calcitriol — Calcitriol is a form of vitamin D given twice daily (BID)
  Other Names: 1,25-dihydroxyvitamin D3
  Arms: Calcitriol 0.25 mcg

SUMMARY:
Men with infertility and normal hormone levels have few options for fertility treatment. Previous research work has suggested that men with infertility may have low levels of the active form of Vitamin A, called retinoic acid, in their testes. We think that giving men with low sperm counts retinoic acid may increase their sperm counts and improve their chances of fathering a pregnancy. We want to see if retinoic acid administration over twenty weeks can increase sperm production and help infertile men become fathers without the need for In vitro fertilization (IVF) and/or intracytoplasmic sperm injection (ICSI). We also want to see if adding calcitriol with retinoic acid will improve sperm motility in a sub-set of subjects.

DETAILED DESCRIPTION:
This is a 20 week, unblinded, two-arm pilot study to determine the impact of therapy with 13-cis retinoic acid and calcitriol on sperm indices in infertile men. Twenty infertile men, ages 21-60 with abnormal sperm analyses will be enrolled for 20-week and given 20 mg 13-cis retinoic acid, twice daily. Subjects#11-#20 will also be administered calcitriol to see if adding calcitriol with Accutane will improve sperm motility. All subjects will be closely followed for side effects related to treatment. The impact of treatment on indices of spermatogenesis will be determined by monthly seminal fluid analyses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be infertile men (no pregnancy with partner with normal cycles and normal hysterosalpingogram despite >1 year of unprotected intercourse).
* Abnormal sperm analyses with a total, motile sperm count of less than 10 million sperm as assessed by semen analysis on two occasions separated by one week.
* In the opinion of the investigator, is able to comply with the protocol, understand and sign an informed consent and HIPAA (Health Insurance Portability and Accountability Act ) form.

Exclusion Criteria:

* Men participating in another clinical trial
* Men not living in the catchment area of the clinic
* Clinically significant abnormal findings at screening
* Known genetic infertility (e.g. Klinefelter syndrome or Y-chromosome microdeletions),
* Hypogonadotropic hypogonadism (that might respond to gonadotropin injections),
* The use of anabolic steroids, illicit drugs, or the consumption of more than 4 alcoholic beverages daily
* Severe mental health problems requiring medications
* Current therapy with retinoic acid (e.g. Accutane) or vitamin A.
* Score of greater than 15 on the Patient health questionnaire (PHQ9).
* Abnormal serum chemistry values according to local laboratory normal values which indicate liver or kidney dysfunction. Other abnormal lab values may also be exclusionary, at the discretion of the investigator
* Men with a personal history of serious psychiatric disorders
* Men currently receiving tetracycline containing medications
* Men currently receiving phenytoin
* Men with a history of inflammatory bowel disease
* Men with a history of bone disease
* Men who have used isotretinoin within eight weeks of the start of dosing
* Men with elevated serum triglycerides

Ages: 21 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-08; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John K Amory, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

REFERENCES:
- [Background] Jequier AM, Holmes SC. Primary testicular disease presenting as azoospermia or oligozoospermia in an infertility clinic. Br J Urol. 1993 Jun;71(6):731-5. doi: 10.1111/j.1464-410x.1993.tb16075.x. PMID 8102079
- [Background] de Kretser DM. Male infertility. Lancet. 1997 Mar 15;349(9054):787-90. doi: 10.1016/s0140-6736(96)08341-9. No abstract available. PMID 9074589
- [Background] Schlegel PN. Nonobstructive azoospermia: a revolutionary surgical approach and results. Semin Reprod Med. 2009 Mar;27(2):165-70. doi: 10.1055/s-0029-1202305. Epub 2009 Feb 26. PMID 19247918
- [Background] Napoli JL. Retinoic acid: its biosynthesis and metabolism. Prog Nucleic Acid Res Mol Biol. 1999;63:139-88. doi: 10.1016/s0079-6603(08)60722-9. PMID 10506831
- [Background] Center for Disease Control. Infertility Facts,m accessed at http://www.ede.gov/nchs/fastats/fertile.htm (June 3, 2013)
- [Background] Doyle TJ, Braun KW, McLean DJ, Wright RW, Griswold MD, Kim KH. Potential functions of retinoic acid receptor A in Sertoli cells and germ cells during spermatogenesis. Ann N Y Acad Sci. 2007 Dec;1120:114-30. doi: 10.1196/annals.1411.008. Epub 2007 Sep 28. PMID 17905941
- [Background] Koubova J, Menke DB, Zhou Q, Capel B, Griswold MD, Page DC. Retinoic acid regulates sex-specific timing of meiotic initiation in mice. Proc Natl Acad Sci U S A. 2006 Feb 21;103(8):2474-9. doi: 10.1073/pnas.0510813103. Epub 2006 Feb 6. PMID 16461896
- [Background] Anderson EL, Baltus AE, Roepers-Gajadien HL, Hassold TJ, de Rooij DG, van Pelt AM, Page DC. Stra8 and its inducer, retinoic acid, regulate meiotic initiation in both spermatogenesis and oogenesis in mice. Proc Natl Acad Sci U S A. 2008 Sep 30;105(39):14976-80. doi: 10.1073/pnas.0807297105. Epub 2008 Sep 17. PMID 18799751
- [Background] Chung SS, Wang X, Wolgemuth DJ. Expression of retinoic acid receptor alpha in the germline is essential for proper cellular association and spermiogenesis during spermatogenesis. Development. 2009 Jun;136(12):2091-100. doi: 10.1242/dev.020040. PMID 19465599
- [Background] Dufour JM, Kim KH. Cellular and subcellular localization of six retinoid receptors in rat testis during postnatal development: identification of potential heterodimeric receptors. Biol Reprod. 1999 Nov;61(5):1300-8. doi: 10.1095/biolreprod61.5.1300. PMID 10529278
- [Background] Lohnes D, Kastner P, Dierich A, Mark M, LeMeur M, Chambon P. Function of retinoic acid receptor gamma in the mouse. Cell. 1993 May 21;73(4):643-58. doi: 10.1016/0092-8674(93)90246-m. PMID 8388780
- [Background] Lufkin T, Lohnes D, Mark M, Dierich A, Gorry P, Gaub MP, LeMeur M, Chambon P. High postnatal lethality and testis degeneration in retinoic acid receptor alpha mutant mice. Proc Natl Acad Sci U S A. 1993 Aug 1;90(15):7225-9. doi: 10.1073/pnas.90.15.7225. PMID 8394014
- [Background] Kastner P, Mark M, Leid M, Gansmuller A, Chin W, Grondona JM, Decimo D, Krezel W, Dierich A, Chambon P. Abnormal spermatogenesis in RXR beta mutant mice. Genes Dev. 1996 Jan 1;10(1):80-92. doi: 10.1101/gad.10.1.80. PMID 8557197
- [Background] Ghyselinck NB, Vernet N, Dennefeld C, Giese N, Nau H, Chambon P, Viville S, Mark M. Retinoids and spermatogenesis: lessons from mutant mice lacking the plasma retinol binding protein. Dev Dyn. 2006 Jun;235(6):1608-22. doi: 10.1002/dvdy.20795. PMID 16586441
- [Background] Hoting VE, Schutte B, Schirren C. [Isotretinoin treatment of acne conglobata. Andrologic follow-up]. Fortschr Med. 1992 Aug 20;110(23):427-30. German. PMID 1398387
- [Background] Vogt HJ, Ewers R. [13-cis-Retinoic acid and spermatogenesis. Spermatological and impulse cytophotometric studies]. Hautarzt. 1985 May;36(5):281-6. German. PMID 3159708
- [Background] Torok L, Kadar L, Kasa M. Spermatological investigations in patients treated with etretinate and isotretinoin. Andrologia. 1987 Nov-Dec;19(6):629-33. doi: 10.1111/j.1439-0272.1987.tb01915.x. PMID 3481225
- [Background] Nya-Ngatchou JJ, Arnold SL, Walsh TJ, Muller CH, Page ST, Isoherranen N, Amory JK. Intratesticular 13-cis retinoic acid is lower in men with abnormal semen analyses: a pilot study. Andrology. 2013 Mar;1(2):325-31. doi: 10.1111/j.2047-2927.2012.00033.x. Epub 2012 Nov 29. PMID 23413144
- [Background] WHO Laboratory Manual for the Examination of Human Semen and Sperm-Cervical Mucus Interaction
- [Background] Christiansen C, Christensen MS, Rodbro P, Hagen C, Transbol I. Effect of 1,25-dihydroxy-vitamin D3 in itself or combined with hormone treatment in preventing postmenopausal osteoporosis. Eur J Clin Invest. 1981 Aug;11(4):305-9. doi: 10.1111/j.1365-2362.1981.tb02121.x. PMID 6795047
- [Background] Riggs BL, Nelson KI. Effect of long term treatment with calcitriol on calcium absorption and mineral metabolism in postmenopausal osteoporosis. J Clin Endocrinol Metab. 1985 Sep;61(3):457-61. doi: 10.1210/jcem-61-3-457. PMID 3926808
- [Background] Falch JA, Odegaard OR, Finnanger AM, Matheson I. Postmenopausal osteoporosis: no effect of three years treatment with 1,25-dihydroxycholecalciferol. Acta Med Scand. 1987;221(2):199-204. doi: 10.1111/j.0954-6820.1987.tb01267.x. PMID 3035879
- [Background] Caniggia A, Nuti R, Lore F, Martini G, Turchetti V, Righi G. Long-term treatment with calcitriol in postmenopausal osteoporosis. Metabolism. 1990 Apr;39(4 Suppl 1):43-9. doi: 10.1016/0026-0495(90)90272-e. PMID 2325571
- [Background] Ott SM, Chesnut CH 3rd. Calcitriol treatment is not effective in postmenopausal osteoporosis. Ann Intern Med. 1989 Feb 15;110(4):267-74. doi: 10.7326/0003-4819-110-4-267. PMID 2913914
- [Background] Gallagher JC, Fowler SE, Detter JR, Sherman SS. Combination treatment with estrogen and calcitriol in the prevention of age-related bone loss. J Clin Endocrinol Metab. 2001 Aug;86(8):3618-28. doi: 10.1210/jcem.86.8.7703. PMID 11502787

RESULTS

PARTICIPANT FLOW:
Groups:
- 13-cis Retinoic Acid + Oral Calcitriol: 20 mg 13-cis retinoic acid twice daily (BID) with meals for two weeks + oral calcitriol 0.25 mcg BID
- 13-cis Retinoic Acid: 20 mg 13-cis retinoic acid twice daily (BID) with meals for 20 weeks
Period: Overall Study
Arm/Group | 13-cis Retinoic Acid + Oral Calcitriol | 13-cis Retinoic Acid
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Sixteen men completed all study procedures, and three men discontinued treatment early.
Groups:
- 13-cis Retinoic Acid + Calcitriol 0.25 mcg: oral calcitriol 025 mcg BID subjects 11-20 for 20 weeks
  Calcitriol: Calcitriol is a form of vitamin D given twice daily (BID)
- Total: Total of all reporting groups
Arm/Group | 13-cis Retinoic Acid | 13-cis Retinoic Acid + Calcitriol 0.25 mcg | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (5.32) | 34 (3.4) | 34.61 (4.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 10 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 9 | 19
  Asian | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Millions of Sperm Per Ejaculate
Description: Millions of sperm per ejaculate in men treated with 13-cis retinoic acid
Time Frame: Up to 20-weeks
Population: First 10 men received isotretinoin alone, next 10 men received both isotretinoin and calcitriol
Measure: Median (Inter-Quartile Range); unit: Millions of sperm per ejaculate
Arm/Group | 13-cis Retinoic Acid | Calcitriol 0.25 mcg
Number analyzed (Participants) | 10 | 10
Millions of sperm per ejaculate | 2.5 [0.1 to 5.9] | 3.8 [2.1 to 13.0]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | 13-cis Retinoic Acid + Oral Calcitriol | 13-cis Retinoic Acid
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 13-cis Retinoic Acid + Oral Calcitriol (N=10) | 13-cis Retinoic Acid (N=10)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-10-29): https://cdn.clinicaltrials.gov/large-docs/84/NCT02061384/Prot_SAP_000.pdf
  • Informed Consent Form (2014-01-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT02061384/ICF_001.pdf